CLINICAL TRIAL: NCT04850950
Title: Safety and Efficacy of Tenofovir Alafenamide to Prevent Perinatal Transmission of Hepatitis B (TAF-PPT): A Multicentre, Prospective, Open-label, Randomized Controlled Trial
Brief Title: Tenofovir Alafenamide to Prevent Perinatal Transmission of Hepatitis B
Acronym: TAF-PPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Henan Provincial People's Hospital (Other); The Sixth People's Hospital of Zhengzhou (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shandong Provincial Hospital (Other Government); Luoyang Central Hospital (Other); First Affiliated Hospital of Nanyang Medical College (Other); Sixth People's Hospital of Kaifeng (Unknown); Luohe Central Hospital (Unknown); Xinyang Central Hospital (Other); Yan'an University Affiliated Hospital (Other); Nanyang Central Hospital (Other); Fifth People's Hospital of Anyang (Unknown)
Responsible Party: Principal Investigator, Qing-Lei Zeng, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-KY-0144-002
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis B; Mother-to-Child Transmission; Safety; Efficacy; Hepatitis B Virus; Tenofovir Alafenamide Fumarate
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tablets; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Tenofovir alafenamide fumarate discontinued at delivery date.
  Interventions: Drug: Tenofovir Alafenamide fumarate 25mg Oral Tablet
- Arm 2 (Experimental): Tenofovir alafenamide fumarate discontinued at postpartum month 1.
  Interventions: Drug: Tenofovir Alafenamide fumarate 25mg Oral Tablet

INTERVENTIONS:
Drug: Tenofovir Alafenamide fumarate 25mg Oral Tablet — Tenofovir alafenamide fumarate initiated from the late pregnancy to the delivery date or postpartum month 1.
  Other Names: VEMLIDY®

SUMMARY:
To investigate the safety and efficacy of tenofovir alafenamide (orally 25 mg per day) treated in inactive chronic hepatitis B virus (HBV)-infected pregnant women with high viral load from the late pregnancy until the delivery date or postpartum 1 month.

DETAILED DESCRIPTION:
The investigators intend to include 240 inactive chronic hepatitis B virus (HBV)-infected pregnant women who have an HBV DNA level higher than 200,000 IU per milliliter. Participants will be randomly assigned, in a 1:1 ratio, to receive tenofovir alafenamide (orally 25 mg per day) from the late pregnancy until the delivery date or postpartum 1 month. All the infants will receive standard immunoprophylaxis (100 IU of hepatitis B immunoglobulin and 10 μg of hepatitis B vaccine within 12 hours of birth; the second injection of 10 μg of HBV vaccine will inject at 1 month; and the third dose of 10 μg of HBV vaccine will give at 6 months). The pregnant women and their infants will be followed until postpartum month 7. The primary outcomes are the birth defects and rates of perinatal transmission of HBV. During the prenatal period or the postnatal period up to 7 months of age, cases of a structural defect in newborns or infants were reported as birth defects. The rate of perinatal transmission was defined as the proportion of infants who are positive for hepatitis B surface antigen at 7 months of age. The secondary safety outcomes are the occurrence of maternal or infant adverse events during the study period. Maternal safety evaluations mainly include any adverse events and complications, hepatitis B virologic breakthrough, alanine aminotransferase flare, and so on. Infant' safety profiles mainly included Apgar scores at 1 minute, any abnormal conditions during the study period, and anthropometric indexes at birth and 7 months of age. The secondary efficacy outcomes are the percentages of mothers with an HBV DNA level of less than 200,000 IU per milliliter just before or at delivery, and the hepatitis B e antigen and surface antigen loss or seroconversion in mothers at postpartum month 7.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age of more than 30 weeks;
2. Had chronic hepatitis B virus (HBV) infection;
3. HBV DNA > 200,000 IU/ml;
4. Consecutively normal levels of alanine aminotransferase (< 40 U/L) and total bilirubin (< 17.1 μmol/L);
5. Willing and able to provide written informed consent and adhere to the trial protocol.

Exclusion Criteria:

1. Previous treatment to reduce alanine aminotransferase and total bilirubin levels;
2. Previous antiviral treatment for HBV infection (except when antiviral agents were administered for the prevention of perinatal transmission during a previous pregnancy and discontinued more than 6 months before the current pregnancy);
3. Coinfection with hepatitis C, D, E, or human immunodeficiency virus;
4. Previous or current evidence of hepatocellular carcinoma, cirrhosis, systemic or other organ disorders;
5. A hemoglobin level of less than 80 g/L;
6. A neutrophil count of less than 1.0 × 10^9/L;
7. An albumin level of less than 30 g/L;
8. Clinical signs of threatened miscarriage;
9. Evidence of fetal deformity by ultrasound examination and other tests;
10. A history of abortion, pregnancy loss, or congenital malformation in a previous pregnancy;
11. A history of genetic disease(s), including the family member(s);
12. Concurrent treatment with other drugs, including but not limited to nephrotoxic drugs, immune modulators, cytotoxic drugs, nonsteroidal antiinflammatory drugs, or steroids.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women.
Enrollment: 240 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth defects. | From prenatal tenofovir alafenamide exposure to the birth and postnatal period up to 7 months of age.
  Structural defect in newborns or infants were reported as birth defects. The monitoring of birth defects was conducted by a clinical examination during each visit, and further clinical imaging or other tests were performed if indicated. The birth defect rate represented the proportion of infants with a defect among all live births.
The rate of perinatal transmission of hepatitis B virus. | At 7 months of age.
  The rate of perinatal transmission was defined as the proportion of infants who are positive for hepatitis B surface antigen at 7 months of age.

SECONDARY OUTCOMES:
Adverse events. | From prenatal tenofovir alafenamide exposure to the delivery (birth) and postnatal period up to 7 months (of age).
  The occurrence of any maternal or infant adverse events.
Alanine aminotransferase flare. | At postpartum month 7.
  Alanine aminotransferase flare was defined as a level greater than 5 or 10 times the upper limit of normal, which was set as 40 U/L according to the Asian-Pacific chronic hepatitis B guideline.
Infants' growth. | At birth and 7 months of age.
  Infant growth was measured by the WHO z scores for age for weight, height, and head circumference.
HBV DNA level. | Immediately before or at delivery.
  Percentage of HBV DNA level of less than 200,000 IU per milliliter for mothers.
Hepatitis B e antigen status. | At postpartum month 7.
  Percentage of hepatitis B e antigen loss or seroconversion for mothers.
Hepatitis B surface antigen status. | At postpartum month 7.
  Percentage of hepatitis B surface antigen loss or seroconversion for mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Qing-Lei Zeng, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

REFERENCES:
- [Derived] Zeng QL, Zhou YH, Dong XP, Zhang JY, Li GM, Xu JH, Chen ZM, Song N, Zhang HX, Chen RY, Lv XY, Huang S, Li WZ, Pan YJ, Feng YH, Li ZQ, Zhang GF, Lin WB, Zhang GQ, Li GT, Li W, Zeng YL, Zhang DW, Cui GL, Lv J, Liu YM, Liang HX, Sun CY, Wang FS, Yu ZJ. Expected 8-Week Prenatal vs 12-Week Perinatal Tenofovir Alafenamide Prophylaxis to Prevent Mother-to-Child Transmission of Hepatitis B Virus: A Multicenter, Prospective, Open-Label, Randomized Controlled Trial. Am J Gastroenterol. 2025 May 1;120(5):1045-1056. doi: 10.14309/ajg.0000000000003122. Epub 2024 Oct 9. PMID 39382852